CLINICAL TRIAL: NCT03840928
Title: PatientSpot Formerly Known as ArthritisPower
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Global Healthy Living Foundation (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Shilpa Venkatachalam, Director, Patient-Centered Research Operations and Ethical Oversight, Global Healthy Living Foundation
Other Study IDs: GlobalHealthyLivingF
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Fibromyalgia; Gout; Crohn Disease; Juvenile Idiopathic Arthritis; Lupus Erythematosus; Myositis; Osteoarthritis; Osteoporosis; Psoriasis; Psoriatic Arthritis; Scleroderma; Dermatomyositis; Inflammatory Bowel Diseases; Polymyositis; Axial Spondyloarthritis; Diffuse Idiopathic Skeletal Hyperostosis; Polymyalgia Rheumatica; Giant Cell Arteritis; Temporal Arteritis; Wegener; Relapsing Polychondritis; Undifferentiated Connective Tissue Disease; Spinal Cord Injuries; Alzheimer Disease; Amyotrophic Lateral Sclerosis; Ataxia; Bell Palsy; Brain Tumor; Cerebral Aneurysm; Epilepsy; Guillain-Barre Syndrome; Headache; Head Injury; Hydrocephalus; Lumbar Disc Disease; Meningitis; Multiple Sclerosis; Muscular Dystrophy; Neurocutaneous Syndromes; Parkinson Disease; Stroke; Cluster Headache; Tension-Type Headache; Chronic Obstructive Pulmonary Disease; Asthma; Lung Cancer; Cystic Fibrosis; Sleep Apnea; Eczema; Alopecia; Chronic Inflammation; Unstable Angina; Heart Attack; Heart Failure; Arrythmia; Valve Heart Disease; High Blood Pressure; Congenital Heart Disease; Peripheral Arterial Disease; Diabetes; Chronic Liver Disease; Obesity
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Fibromyalgia; Gout; Crohn Disease; Arthritis, Juvenile; Myositis; Osteoarthritis; Osteoporosis; Psoriasis; Arthritis, Psoriatic; Scleroderma, Diffuse; Dermatomyositis; Inflammatory Bowel Diseases; Polymyositis; Axial Spondyloarthritis; Hyperostosis, Diffuse Idiopathic Skeletal; Polymyalgia Rheumatica; Giant Cell Arteritis; Granulomatosis with Polyangiitis; Polychondritis, Relapsing; Undifferentiated Connective Tissue Diseases; Spinal Cord Injuries; Alzheimer Disease; Amyotrophic Lateral Sclerosis; Ataxia; Bell Palsy; Brain Neoplasms; Intracranial Aneurysm; Epilepsy; Guillain-Barre Syndrome; Headache; Craniocerebral Trauma; Hydrocephalus; Intervertebral disc disease; Meningitis; Multiple Sclerosis; Muscular Dystrophies; Neurocutaneous Syndromes; Parkinson Disease; Stroke; Cluster Headache; Tension-Type Headache; Pulmonary Disease, Chronic Obstructive; Asthma; Lung Neoplasms; Cystic Fibrosis; Sleep Apnea Syndromes; Eczema; Alopecia; Angina, Unstable; Myocardial Infarction; Heart Failure; Arrhythmias, Cardiac; Heart Valve Diseases; Hypertension; Heart Defects, Congenital; Peripheral Arterial Disease; Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (13):
- Ankylosing Spondylitis
- Fibromyalgia
- Gout
- Crohn's-related Arthritis
- Juvenile Idiopathic Arthritis
- Lupus
- Myositis
- Osteoarthritis
- Osteoporosis
- Psoriasis
- Psoriatic Arthritis
- Rheumatoid Arthritis
- Scleroderma

SUMMARY:
Patient Power is a patient research network and database (registry) to collect prospective information about demographics, self-reported diagnoses and medications, and willingness to participate in research from participants with rheumatoid arthritis (RA), spondyloarthritis (SpA), other musculoskeletal conditions, chronic neurological conditions like migraine, chronic pulmonary conditions like Chronic Obstructive Pulmonary Disease (COPD), asthma, autoimmune dermatological conditions such as psoriasis, and other chronic inflammatory or immune-mediated conditions. In addition, since patients with chronic conditions often have other co-morbidities like cardiovascular health and obesity-related metabolic disorders, these conditions will also be included. Participants will provide information from their smartphones or personal computers. The information will be used by researchers and clinicians to help patients and their providers make better, more informed decisions about treatment of chronic conditions.

DETAILED DESCRIPTION:
Patient Power is a patient research network and database (registry) to collect prospective information about demographics, self-reported diagnoses and medications, and willingness to participate in research from participants with rheumatoid arthritis (RA), spondyloarthritis (SpA), other musculoskeletal conditions, chronic neurological conditions like migraine, chronic pulmonary conditions like Chronic Obstructive Pulmonary Disease (COPD), asthma, autoimmune dermatological conditions such as psoriasis, and other chronic inflammatory or immune-mediated conditions. In addition, since patients with chronic conditions often have other co-morbidities like cardiovascular health and obesity-related metabolic disorders, these conditions will also be included. Participants will provide information from their smartphones or personal computers. The information will be used by researchers and clinicians to help patients and their providers make better, more informed decisions about treatment of chronic conditions.

We have established a governance structure with highly engaged patients and stakeholders who will serve on a Patient Governor Group (PGG) and Research Advisory Board (RAB) to ensure Patient Power participant privacy and transparency about research activities. Online tools and a mobile application at me securely capture patient data. The software tools built include real-time connection to the adaptive version of NIH Patient Reported Outcomes Measurement Information System (PROMIS) instruments capturing patient reported data that minimizes participant burden and allows participants to immediately view their scores if they choose. The Patient Power App runs on both web browsers and smartphones with data stored in the Amazon Web Services (AWS) cloud, not on a participant's smartphone or browser. The App has four key design pillars: (1) Patient engagement, community integration and education by incorporating GHLF bloggers and chronic disease news and social media engagement to the app for education, support and research findings to be shared directly and immediately with those living with registry-eligible chronic conditions; (2) Personal longitudinal health and medication tracking by providing participants' access to their actively contributed patient reported outcome (PRO) and other health-related data (e.g. current and past medications). We will use messaging to encourage participants to regularly update their information, including medication information. For example, we may remind participants to contribute their medication information with the following message: "You don't have any active medications. You can record your medications in Patient Power. By adding your active medications, you will be able to see how your symptoms have changed since starting a new medication. Click here to start entering medications". (3) Health care decision making by allowing App users to share health tracking reports at their discretion with their providers or caregivers; and (4) Research opportunities by providing a platform where an array of new research opportunities can be browsed by participants to combat chronic diseases. The combination of solid governance structure with well-developed policies and procedures, engaged patient community, collaborative relationships with many research partners and our innovatively convenient and mobile approach to data collection make Patient Power a unique and powerful patient-led initiative in chronic disease research.

ELIGIBILITY:
Inclusion Criteria:

* Self-report that a physician has given a diagnosis of a chronic condition listed in the registry.
* The Registry is only intended at this time for residents of the United States and United States territories and Canada who are nineteen (19) years or older (for Puerto Rico residents, you must be 21 years or older to participate).

Exclusion Criteria

• Under 19 years old

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be derived from the population of people who indicate that they have been diagnosed by a physician with a chronic condition. al conditions will be invited to join the ArthritisPower research registry and download the PatientSpot App.
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain Interference (PROMIS) | 7 days
Fatigue (PROMIS) | 7 days
Sleep Disturbance (PROMIS) | 7 days
Physical Function (PROMIS) | 7 days
RAPID-3 (MD-HAQ with visual analogue scale for pain and patient global measure for overall health) | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Global Healthy Living Foundation, Upper Nyack, New York, United States